CLINICAL TRIAL: NCT02002208
Title: A Study of the Effect of OC000459 on Signs and Symptoms in Subjects With Moderate to Severe Atopic Dermatitis: A Randomised Double Blind Placebo Controlled Parallel Group Study
Brief Title: Effect of OC000459 on Moderate to Severe Atopic Dermatitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Atopix Therapeutics, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OC000459/017/13
Record Dates: First submitted 2013-11-26; First posted 2013-12-05 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2018-03-26 (Actual); Status verified 2018-02

CONDITIONS: Atopic Dermatitis
MeSH Terms: conditions — Dermatitis, Atopic | interventions — (5-fluoro-2-methyl-3-quinolin-2-ylmethylindo-1-yl)acetic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- OC000459 Tablets (Experimental): 50 mg orally once a day
  Interventions: Drug: OC000459
- Placebo Tablets (Placebo Comparator): Orally once a day
  Interventions: Drug: OC000459

INTERVENTIONS:
Drug: OC000459 — Oral CRTH2 antagonist
  Other Names: timapiprant

SUMMARY:
The purpose of this study is to determine whether OC000459 is in reducing disease severity and preventing flares in people with moderate to severe atopic dermatitis (AD).

DETAILED DESCRIPTION:
The study will include patients with a Th2 high eosinophilic phenotype who typically have more severe disease and are prone to flare.

ELIGIBILITY:
Inclusion Criteria:

1. Atopic dermatitis as defined by a score of at least 9 on the Nottingham Eczema Severity Score, stratified into moderate (score 9 to 11 inclusive) and severe (score 12 to 15 inclusive) disease.
2. Fully documented history of the use of topical corticosteroids (TCS) and/or topical calcineurin inhibitors (TCI). Subjects without a fully documented history will be excluded from the study.
3. Male and female subjects with moderate to severe atopic dermatitis treated with by TCS and/or TCI (with or without emollients) at the time of screening and over the previous month.
4. Subjects must have had at least 1 AD flare in the previous 6 months.

Exclusion Criteria:

1. Receipt of any forbidden medication including over the counter preparations and herbal medicines within 14 days of the first dosing day with the exception of paracetamol up to a maximum of 2g daily.
2. Use of systemic steroids within 4 weeks of the screening visit, light therapy or immunosuppressants within 2 months of the screening visit.
3. Use of NSAIDs.
4. Subjects initially diagnosed with AD aged 2 years or over will be excluded unless they have either coexisting or a history of asthma and/or allergic rhinoconjunctivitis.
5. Subjects with contact dermatitis will be excluded.
6. Subjects with acute skin infection or acute disease flares. Subjects with active flares during the screening to randomisation period (visits 1 to 2) may be managed according to normal clinical practice and be rescreened once their flares are no longer active.

   -

Ages: 18 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 142 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Cork, MB, Principal Investigator — University of Sheffield
Locations (1):
- University of Sheffield, Sheffield, United Kingdom

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 142 patients were randomised. One patient withdrew prior to dosing meaning that there was 141 patients in the safety set. 2 further patients withdrew prior to the first efficacy measurement which means there were 139 patients in the full analysis set.
Groups:
- OC000459 Tablets: 50 mg orally once a day
  OC000459: CRTH2 inhibitor
- Placebo Tablets: Orally once a day
  OC000459: CRTH2 inhibitor
Period: Overall Study
Arm/Group | OC000459 Tablets | Placebo Tablets
Started | 69 | 70
Completed | 32 | 30
Not Completed | 37 | 40

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OC000459 Tablets | Placebo Tablets | Total
Number analyzed (Participants) | 69 | 70 | 139
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.6 (8.42) | 30.9 (8.54) | 31.2 (8.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 31 | 60
  Male | 40 | 39 | 79

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Eczema Area and Severity Index (EASI) Compared to Placebo at Week 16
Description: The EASI scoring system uses a defined process to grade the severity of the signs of eczema and the extent affected in four regions of the body: head and neck, trunk, upper extremities and lower extremities. The scale ranges from 0 to 72 and the severity strata for the EASI are as follows: 0 clear; 0.1-1.0 almost clear; 1.1-7.0 mild; 7.1-21.0 =moderate; 21.1-50.0 severe; 50.1-72.0 very severe. When assessing response to therapy a reduction of 7 or more is considered to be clinically meaningful.
Time Frame: EASI was measured at baseline (week 0) and 16 weeks after dosing.
Population: Adjusted mean change from baseline EASI at Week 16
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | OC000459 Tablets | Placebo Tablets
Number analyzed (Participants) | 69 | 70
units on a scale | -3.8 (1.72) | -6.1 (1.71)

2. Secondary Outcome: Rate of Flares
Time Frame: over 16 weeks
Measure: Mean (Standard Deviation); unit: flares
Arm/Group | OC000459 Tablets | Placebo Tablets
Number analyzed (Participants) | 69 | 70
flares | 2.879 (2.8679) | 2.646 (4.7922)

ADVERSE EVENTS:
Time Frame: Up to 6 months
Description: Standardised coding using MedDRA
Arm/Group | OC000459 Tablets | Placebo Tablets
Serious Adverse Events (participants affected / at risk) | 2/70 | 6/71
Other Adverse Events (participants affected / at risk) | 52/70 | 47/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | OC000459 Tablets (N=70) | Placebo Tablets (N=71)
Worsening atopic dermatitis (Skin and subcutaneous tissue disorders) | 1 | 3
Staphylococcal infection (Infections and infestations) | 0 | 1
Anaphylaxis (Immune system disorders) | 0 | 1 — Anaphylaxis due to peanut allergy
ECG abnormality (Investigations) | 0 | 1
Gastroenteritis (Gastrointestinal disorders) | 0 | 1
Solitary Plasmacytoma (Blood and lymphatic system disorders) | 1 | 0 — Event occurred 6 months after last dose of study medication
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | OC000459 Tablets (N=70) | Placebo Tablets (N=71)
Headache (Nervous system disorders) | 15 | 15
Nasopharyngitis (Infections and infestations) | 9 | 15
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 4
Herpes simplex (Infections and infestations) | 4 | 2
Nausea (Gastrointestinal disorders) | 3 | 4
Tooth ache (Gastrointestinal disorders) | 0 | 3
Fatigue (General disorders) | 0 | 3
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 3
Cystitis (Infections and infestations) | 2 | 0
Ear infection (Infections and infestations) | 0 | 2
Rash pustular (Infections and infestations) | 2 | 0
Tonsillitis (Infections and infestations) | 0 | 2
Disturbance in attention (Nervous system disorders) | 0 | 2
Dizziness (Nervous system disorders) | 0 | 2
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 6 | 5
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Conjunctivitis (Eye disorders) | 2 | 1
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 2
Chest pain (General disorders) | 2 | 0
Influenza like illness (General disorders) | 2 | 0
Insomnia (Psychiatric disorders) | 2 | 0
Panic attack (Psychiatric disorders) | 0 | 2
Sleep disorder (Psychiatric disorders) | 0 | 2
Food allergy (Immune system disorders) | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No